CLINICAL TRIAL: NCT02508532
Title: A Phase 1 Study of BLU-285 in Patients With Gastrointestinal Stromal Tumors (GIST) and Other Relapsed and Refractory Solid Tumors
Brief Title: (NAVIGATOR) Study of BLU-285 in Patients With Gastrointestinal Stromal Tumors (GIST) and Other Relapsed and Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-1101
Expanded Access: NCT03862885 (Approved for marketing)
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2021-07

CONDITIONS: Gastrointestinal Stromal Tumors (GIST); Other Relapsed or Refractory Solid Tumors
Keywords: 2L GIST; GIST second line; GIST gleevec; GIST imatinib; Second-line GIST clinical trial; BLU-285; BLU 285; BLUE-285; BLUE 285; Avapritinib; GIST imatinib relapse; GIST gleevec relapse; GIST KIT; GIST relapse; GIST refractory; GIST imatinib intolerance; GIST TKI treatment; GIST tyrosine kinase inhibitor treatment; GIST TKI; GIST tyrosine kinase inhibitor; Advanced GIST; GIST mutations; GIST treatments; Blueprint GIST; Relapsed GIST clinical trial; Refractory GIST clinical trial; KIT-mutant GIST; cancer gist; gastrointestinal stromal tumor; gist cancer; PDGFRA
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — avapritinib

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Dose Expansion
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part 1 Avapritinib (formerly BLU-285) 30 mg QD (Experimental): Part 1: Patients received a starting dose of 30 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 60 mg QD (Experimental): Part 1: Patients received a starting dose of 60 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 90 mg QD (Experimental): Part 1: Patients received a starting dose of 90 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 135 mg QD (Experimental): Part 1: Patients received a starting dose of 135 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 200 mg QD (Experimental): Part 1: Patients received a starting dose of 200 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation. .
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 300 mg QD (Experimental): Part 1: Patients received a starting dose of 300 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation. Patients that received at least one dose of avapritinib were included in the Part 2 analysis.
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 400 mg QD (Experimental): Part 1: Patients received a starting dose of 400 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Patients that received at least one dose of avapritinib were included in the Part 2 analysis.
  Interventions: Drug: Avapritinib
- Part 1 Avapritinib (formerly BLU-285) 600 mg QD (Experimental): Part 1: Patients received a starting dose of 600 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Interventions: Drug: Avapritinib
- Part 1 and Part 2 Avapritinib (formerly BLU-285) 300 mg or 400 mg QD (Experimental): Part 1 and Part 2: Patients enrolled in Part 1 and Part 2 at a starting dose of 300 or 400 mg QD were included in the Part1/Part 2 safety and efficacy analysis.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — avapritinib tablets
  Other Names: BLU-285

SUMMARY:
This is a Phase 1, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antineoplastic activity of avapritinib (formerly BLU-285), administered orally (PO), in adult patients with unresectable GIST or other relapsed or refractory solid tumors. The study consists of 2 parts, a dose-escalation part (Part 1) and an expansion part (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* For Part 1: Histologically- or cytologically-confirmed diagnosis of unresectable GIST or another advanced solid tumor. Patients with unresectable GIST must have disease that has progressed following imatinib and at least 1 of the following: sunitinib, regorafenib, sorafenib, dasatinib, pazopanib or an experimental kinase-inhibitor agent, or disease with a D842 mutation in the PDGFRα gene. Patients with an advanced solid tumor other than GIST must have relapsed or refractory disease without an available effective therapy.

OR For Part 2:

* Group 1: Patients must have a confirmed diagnosis of unresectable GIST that has progressed following imatinib and at least 1 of the following: sunitinib, regorafenib, sorafenib, dasatinib, pazopanib, or an experimental kinase-inhibitor agent, and the patient does not have a D842V mutation in PDGFRα.
* Group 2: Patients must have a confirmed diagnosis of unresectable GIST with a D842V mutation in the PDGFRα gene. The PDGFRα mutation will be identified by local or central assessment, either in an archival tissue sample or a new tumor biopsy obtained prior to treatment with avapritinib.
* Group 3: Patients must have a confirmed diagnosis of unresectable GIST that has progressed and/or patients must have experienced intolerance to imatinib and not received additional kinase-inhibitor therapy. Patients must not have a known D842V mutation in PDGFRα.
* Groups 1, 2 and 3: At least 1 measurable lesion defined by mRECIST 1.1 for patients with GIST.
* Groups 1 and 2: A tumor sample (archival tissue or a new tumor biopsy) has been submitted for mutational testing.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* QT interval corrected using Fridericia's formula (QTcF) >450 milliseconds
* Platelet count <90,000/mL
* Absolute neutrophil count <1000/mL
* Hemoglobin <9 g/dL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 x the upper limit of normal (ULN) if no hepatic metastases are present; >5 × ULN if hepatic metastases are present
* Total bilirubin >1.5 × ULN; >3 × ULN with direct bilirubin, >1.5 × ULN in the presence of Gilbert's Disease
* Estimated (Cockroft-Gault formula) or measured creatinine clearance <40 mL/min Brain malignancy or metastases to the brain
* History of a seizure disorder or requirement for anti-seizure medication
* Group 3: Patients known to be KIT wild type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2021-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (9):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - Sarcoma Oncology Center, Santa Monica, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Cancer Treatment Centers of America, Atlanta, Georgia
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Leuven Cancer Institute University Hospitals Leuven, Leuven, Belgium
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Paris
- University of Duisburg-Essen, Essen, Germany
- Fondazione IRCCS - Istituto Nazinale dei Tumori, Milan, Italy
- Erasmus MC Cancer Institute, Rotterdam, Netherlands
- Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie w Warszawie, Warsaw, Poland
- Asan Medical Center, Seoul, South Korea
- Vall d' Hebron Institute of Oncology (VHIO), Barcelona, Spain
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- [Derived] Kang YK, George S, Jones RL, Rutkowski P, Shen L, Mir O, Patel S, Zhou Y, von Mehren M, Hohenberger P, Villalobos V, Brahmi M, Tap WD, Trent J, Pantaleo MA, Schoffski P, He K, Hew P, Newberry K, Roche M, Heinrich MC, Bauer S. Avapritinib Versus Regorafenib in Locally Advanced Unresectable or Metastatic GI Stromal Tumor: A Randomized, Open-Label Phase III Study. J Clin Oncol. 2021 Oct 1;39(28):3128-3139. doi: 10.1200/JCO.21.00217. Epub 2021 Aug 3. PMID 34343033
- [Derived] von Mehren M, Heinrich MC, Shi H, Iannazzo S, Mankoski R, Dimitrijevic S, Hoehn G, Chiroli S, George S. Clinical efficacy comparison of avapritinib with other tyrosine kinase inhibitors in gastrointestinal stromal tumors with PDGFRA D842V mutation: a retrospective analysis of clinical trial and real-world data. BMC Cancer. 2021 Mar 19;21(1):291. doi: 10.1186/s12885-021-08013-1. PMID 33740926
- [Derived] Jones RL, Serrano C, von Mehren M, George S, Heinrich MC, Kang YK, Schoffski P, Cassier PA, Mir O, Chawla SP, Eskens FALM, Rutkowski P, Tap WD, Zhou T, Roche M, Bauer S. Avapritinib in unresectable or metastatic PDGFRA D842V-mutant gastrointestinal stromal tumours: Long-term efficacy and safety data from the NAVIGATOR phase I trial. Eur J Cancer. 2021 Mar;145:132-142. doi: 10.1016/j.ejca.2020.12.008. Epub 2021 Jan 16. PMID 33465704
- [Derived] Joseph CP, Abaricia SN, Angelis MA, Polson K, Jones RL, Kang YK, Riedel RF, Schoffski P, Serrano C, Trent J, Tetzlaff ED, Si TD, Zhou T, Doyle A, Bauer S, Roche M, Havnaer T. Optimal Avapritinib Treatment Strategies for Patients with Metastatic or Unresectable Gastrointestinal Stromal Tumors. Oncologist. 2021 Apr;26(4):e622-e631. doi: 10.1002/onco.13632. Epub 2021 Jan 5. PMID 33301227
- [Derived] Heinrich MC, Jones RL, von Mehren M, Schoffski P, Serrano C, Kang YK, Cassier PA, Mir O, Eskens F, Tap WD, Rutkowski P, Chawla SP, Trent J, Tugnait M, Evans EK, Lauz T, Zhou T, Roche M, Wolf BB, Bauer S, George S. Avapritinib in advanced PDGFRA D842V-mutant gastrointestinal stromal tumour (NAVIGATOR): a multicentre, open-label, phase 1 trial. Lancet Oncol. 2020 Jul;21(7):935-946. doi: 10.1016/S1470-2045(20)30269-2. PMID 32615108
- [Derived] Gebreyohannes YK, Wozniak A, Zhai ME, Wellens J, Cornillie J, Vanleeuw U, Evans E, Gardino AK, Lengauer C, Debiec-Rychter M, Sciot R, Schoffski P. Robust Activity of Avapritinib, Potent and Highly Selective Inhibitor of Mutated KIT, in Patient-derived Xenograft Models of Gastrointestinal Stromal Tumors. Clin Cancer Res. 2019 Jan 15;25(2):609-618. doi: 10.1158/1078-0432.CCR-18-1858. Epub 2018 Oct 1. PMID 30274985

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD: Part 1: Patients received a starting dose of 30 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD: Part 1: Patients received a starting dose of 60 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD: Part 1: Patients received a starting dose of 90 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD: Part 1: Patients received a starting dose of 135 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD: Part 1: Patients received a starting dose of 200 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation. .
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 300 mg QD: Part 1: Patients received a starting dose of 300 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 400 mg QD: Part 1: Patients received a starting dose of 400 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD: Part 1: Patients received a starting dose of 600 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD: Part 1 and Part 2: Patients enrolled in Part 1 and Part 2 at a starting dose of 300 or 400 mg QD were included in the Part1/Part 2 safety and efficacy analysis.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
Period: Part 1 - Dose Determining Period
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 300 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 400 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD
Started | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 3 | 0 (This group includes patients enrolled in Part 1 and Part 2 at a starting dose of 300 or 400 mg QD. This group was not used to determine the MTD in Part 1)
Patients From Part 1 Included in the Part 2 Analyses | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — did not complete >21 days of treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Not Evaluable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 2 - Treatment
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 300 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 400 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD
Started | 0 (These patients are not included in Part 2 analyses) | 0 (These patients are not included in Part 2 analyses) | 0 (These patients are not included in Part 2 analyses) | 0 (These patients are not included in Part 2 analyses) | 0 (These patients are not included in Part 2 analyses) | 0 (Part 1 Only: 6 Patients from this group are included in the 300 or 400 mg QD group.) | 0 (Part 1 Only: 7 Patients from this group are included in the 300 or 400 mg QD group.) | 0 (These patients are not included in Part 2 analyses) | 217 (Includes 13 patients enrolled in Part 1 at a starting dose of 300 mg (n = 6) or 400 mg (n = 7) QD.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 217
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 118
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 49
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Not completed — Administrative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Period: Part 1 and Part 2 End of Study
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 300 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 400 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD
Started | 6 | 6 | 6 | 6 | 6 | 0 (These 6 patients are included in the 300 or 400 mg QD dose group) | 0 (These 7 patients are included in the 300 or 400 mg QD dose group) | 3 | 217 (Includes 13 patients enrolled in Part 1 at a starting dose of 300 mg (n = 6) or 400 mg (n = 7) QD.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 3 | 217
Not completed — Disease Progression | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 4 | 2 | 4 | 3 | 0 | 0 | 1 | 111
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 8
Not completed — Initiation of another therapy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 2 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 68

BASELINE CHARACTERISTICS:
Groups:
- Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 mg or 400 mg QD: Part 1 and Part 2: Patients enrolled in Part 1 and Part 2 at a starting dose of 300 or 400 mg QD were included in the Part1/Part 2 safety and efficacy analysis.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Includes 13 patients from Part 1
- Total: Total of all reporting groups
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD | Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 mg or 400 mg QD | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 3 | 217 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (12.21) | 60.2 (6.77) | 60.2 (11.84) | 61.5 (10.05) | 61.7 (8.31) | 48.3 (20.82) | 59.4 (11.00) | 59.4 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 0 | 3 | 1 | 84 | 96
  Male | 2 | 3 | 5 | 6 | 3 | 2 | 133 | 154
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 10 | 12
  White | 5 | 6 | 4 | 5 | 4 | 3 | 154 | 181
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2 | 0 | 28 | 32
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 0 | 1 | 1 | 1 | 0 | 13 | 16
  France | 0 | 0 | 1 | 1 | 2 | 0 | 20 | 24
  Germany | 1 | 2 | 0 | 1 | 0 | 0 | 14 | 18
  Netherlands | 0 | 0 | 1 | 0 | 0 | 0 | 11 | 12
  Poland | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
  South Korea | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 17
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11
  United Kingdom | 1 | 0 | 3 | 0 | 0 | 1 | 23 | 28
  United States | 4 | 4 | 0 | 3 | 3 | 2 | 100 | 116
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Population: Body Mass Index was only calculated for patients with both a height and weight measurement at Baseline
  kg/m2
    number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 3 | 198 | 228
    (all) | 24.78 (4.22) | 31.61 (8.63) | 28.33 (3.76) | 23.78 (2.71) | 24.63 (5.16) | 27.15 (4.54) | 25.98 (6.22) | 26.09 (6.15)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Avapritinib
Description: Patients with event(s) of dose-limiting toxicity
Time Frame: Cycle 1 (28 days) of treatment
Population: Patients that completed Part 1 or had a DLT
Measure: Number; unit: patients with event(s) of dose-limiting
Groups:
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 300 mg QD: Part 1: Patients received a starting dose of 300 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation. Patients that received at least one dose of avapritinib were included in the Part 2 analysis.
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 400 mg QD: Part 1: Patients received a starting dose of 400 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
  Patients that received at least one dose of avapritinib were included in the Part 2 analysis.
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 300 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 400 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 2
patients with event(s) of dose-limiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Parts 1 and 2: Number of Patients With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: The overall safety profile of the drug was assessed by reviewing the number of patients with AEs, SAEs and other events. There was no formal statistical analysis. Safety assessments continued for the duration of treatment.
Time Frame: AEs were collected from the start of study drug until 30 days after the last dose, SAEs were collected from the date of the informed consent signature until 30 days after the last dose of study drug, up to 5 years
Population: Safety Population - all patients that received at least one dose of avapritinib
Measure: Number; unit: participants
Groups:
- Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 mg or 400 mg QD: Part 1 and Part 2: Patients enrolled in Part 1 and Part 2 at a starting dose of 300 or 400 mg QD were included in the Part1/Part 2 safety and efficacy analysis. 13 patients in this group were enrolled in Part 1
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 mg or 400 mg QD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 3 | 217
participants
  Participants with an Adverse Event | 6 | 6 | 6 | 6 | 6 | 3 | 216
  Participants with a Serious Adverse Event | 3 | 4 | 5 | 5 | 5 | 3 | 140

3. Primary Outcome: Part 2: Objective Response Rate (ORR) Determined by Central Radiology Assessment Per mRECIST, Version 1.1
Description: To evaluate objective response rate (ORR) determined by central radiology assessment per mRECIST, version 1.1 in patients with advanced GIST treated with avapritinib. A complete response per modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) is defined as complete disappearance of all target lesions. A partial response is defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters. Overall Response (OR) = CR + PR
Time Frame: Tumor assessments were performed at screening, Cycle 3 Day 1, then every 2 cycles through Cycle 13, then every 3 cycles thereafter up to approximately 4 years. Each cycle is 28 days.
Population: patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg, including 13 patients enrolled in Part 1
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a PDGFRA D842V Mutation: Patients with a PDGFRA D842V Mutation, any line of treatment
- 2L Patients Without a PDGFRA D842V Mutation: Patients that do not have a PDGFRA D842V mutation and have received 1 prior line of therapy
- 3L Patients Without a PDGFRA D842V Mutation: Patients that do not have a PDGFRA D842V mutation and have had 2 or more prior lines of therapy
Arm/Group | Patients With a PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 38 | 50 | 128
Participants
  Responder | 36 | 10 | 20
  Non-Responder | 2 | 40 | 108

4. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax)
Description: Maximum plasma drug concentration (Cmax) following a single dose of avapritinib
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available samples for PK
Measure: Median (Standard Deviation); unit: ng/mL
Groups:
- Part 1 Avapritinib (Formerly BLU-285) 300 mg QD: Part 1 and Part 2: Patients received a starting dose of 300 mg QD. Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Part 1 Avapritinib (Formerly BLU-285) 400 mg QD: Part 1 and Part 2: Patients received a starting dose of 400 mg QD. Patients received avapritinib in continuous 28 day cycles until discontinuation.
Arm/Group | Part 1 Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 113 | 50
ng/mL | 305 (153) | 343 (181)

5. Secondary Outcome: Time to Maximum Plasma Drug Concentration (Tmax)
Description: Cycle 1 Day 1 PK time to maximum plasma drug concentration (Tmax)
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 and Part 2 with available samples for PK
Measure: Median (Full Range); unit: hours
Groups:
- Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD: Part 1 and Part 2: Patients received a starting dose of 300 mg QD. Patients received avapritinib in continuous 28 day cycles until discontinuation.
- Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD: Part 1 and Part 2: Patients received a starting dose of 400 mg QD. Patients received avapritinib in continuous 28 day cycles until discontinuation.
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 113 | 50
hours | 4.0 [0.98 to 23.5] | 4.02 [1.97 to 24.0]

6. Secondary Outcome: Plasma Drug Concentration at 24 Hours Postdose Prior to the Next Daily Dose (C24)
Description: Plasma drug concentration at 24 hours postdose prior to the next daily dose (C24) following a single dose of avapritinib
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg QD and available PK samples
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 36 | 19
ng/mL | 134 (49.4) | 185 (80.2)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours (AUC 0-24)
Description: Area under the plasma concentration-time curve from time 0 to 24 hours (AUC 0-24) following a single dose of avapritinib
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg QD and available PK samples
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 36 | 19
h*ng/mL | 4510 (1760) | 5310 (2080)

8. Secondary Outcome: Apparent Oral Clearance Unadjusted for Bioavailability (CL/F)
Description: Apparent oral clearance unadjusted for bioavailability (CL/F) following a single dose of avapritinib
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg QD and available PK samples
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 23 | 8
L/h | 31.5 (15.2) | 29.9 (20.1)

9. Secondary Outcome: Apparent Volume of Distribution, Unadjusted for Bioavailability (Vz/F)
Description: Apparent volume of distribution, unadjusted for bioavailability (Vz/F) following a single dose of avapritinib
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available PK samples
Measure: Mean (Standard Error); unit: L
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 23 | 8
L | 1310 (676) | 1340 (597)

10. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: Terminal elimination half-life (t1/2) following a single dose of avapritinib
Time Frame: Cycle 1 Day 1
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg QD and available PK samples
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 23 | 8
h | 32.1 (15.6) | 43.5 (28.4)

11. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax) at Steady State
Description: Maximum plasma drug concentration (Cmax) at steady state following 15 days of QD dosing
Time Frame: Cycle 1 Day 15
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available samples for PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 110 | 38
ng/mL | 905 (402) | 1140 (469)

12. Secondary Outcome: Time of Maximal Concentration (Tmax) at Steady State
Description: Time of maximal concentration (Tmax) at steady state following 15 days of QD dosing
Time Frame: Cycle 1 Day 15
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available samples for PK
Measure: Median (Full Range); unit: h
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 110 | 38
h | 4.0 [0.0 to 8.17] | 3.99 [0.5 to 8.0]

13. Secondary Outcome: Plasma Drug Concentration at 24 Hours Postdose Prior to the Next Daily Dose at Steady State (C24,ss)
Description: Plasma Drug Concentration at 24 Hours Postdose Prior to the Next Daily Dose at steady state (C24,ss) following 15 days of QD dosing
Time Frame: Cycle 1 Day 15
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available samples for PK
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 110 | 38
ng/mL | 593 (263) | 760 (343)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dosing Interval at Steady Sate (AUC0-τ,ss) (τ=24 h)
Description: Area under the plasma concentration-time curve over the dosing interval at steady sate (AUC0-τ,ss) (τ=24 h) following 15 days of QD dosing
Time Frame: Cycle 1 Day 15
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available samples for PK
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 110 | 38
h*ng/mL | 16900 (7230) | 21300 (9250)

15. Secondary Outcome: Progression-free Survival Per mRECIST Version 1.1
Description: Progression-free survival is defined as the time in months from the start of treatment to the date of first documented progression or death due to any cause. Progression-free survival determined by central radiological assessment per modified Response Evaluation Criteria in Solid Tumors (mRECIST), version 1.1 in patients with advanced GIST. A progressively growing tumor must meet the following criteria: a) the target lesions must be greater or equal to 2cm in size and be a new GIST active lesion or b) the target lesions must be expanding on at least 2 sequential imaging studies.
Time Frame: as for outcome 3
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg QD
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With a PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 38 | 50 | 128
months | 27.6 [19.5 to NA] — The upper bounds of the confidence interval could not be calculated | 5.5 [2.0 to 9.4] | 3.7 [3.6 to 5.6]

16. Secondary Outcome: Apparent Oral Clearance at Steady State, Unadjusted for Bioavailability (CLss/F)
Description: Apparent oral clearance at steady state, unadjusted for bioavailability (CLss/F) following 15 days of QD dosing
Time Frame: Cycle 1 Day 15
Population: Patients enrolled in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD and available samples for PK
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 300 mg QD | Part 1 and Part 2: Avapritinib (Formerly BLU-285) 400 mg QD
Number analyzed (Participants) | 110 | 38
L/h | 21.8 (12.0) | 22.8 (11.7)

17. Secondary Outcome: Clinical Benefit Rate Determined by Central Radiology Assessment Per mRECIST, Version 1.1
Description: Percent of patients with a complete response, partial response or stable disease lasting more than 16 weeks. A complete response per modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) is defined as complete disappearance of all target lesions. A partial response is defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters. Stable disease is defined as a tumor that does not meet the criteria for progression or for response. A progressively growing tumor must meet the following criteria: a) the target lesions must be greater or equal to 2cm in size and be a new GIST active lesion or b) the target lesions must be expanding on at least 2 sequential imaging studies.
Time Frame: as for outcome 3
Population: patients with a starting dose of 300 or 400 mg QD
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With a PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 38 | 50 | 128
Participants
  Clinical Benefit | 37 | 26 | 51
  No Clinical Benefit | 1 | 24 | 77

18. Secondary Outcome: Response Rate Determined by Central Radiology Assessment Per Choi Criteria
Description: A complete response is defined as complete disappearance of all target lesions. A partial response is ≥10% decrease tumor size at computed tomography (CT) or ≥15% decrease in tumor attenuation at computed tomography (CT) and no new lesions. The response rate is defined as complete response plus partial response.
Time Frame: as for outcome 3
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With a PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 38 | 50 | 128
Participants
  Responder | 37 | 18 | 45
  Non-responder | 1 | 32 | 83

19. Secondary Outcome: Duration of Response Determined by Central Radiology Assessment Per mRECIST, Version 1.1
Description: Duration from time to first documented CR/PR to date of first documented disease progression or death.
  A complete response per modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) is defined as complete disappearance of all target lesions. A partial response is defined as at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters. Overall Response (OR) = CR + PR
Time Frame: as for outcome 3
Population: Patients in Part 1 and Part 2 with a starting dose of 300 or 400 mg QD. Only patients that achieved a CR or PR are included in this analysis
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Patients With PDGFRA D842V Mutation: Patients with a PDGFRA D842V mutation, any line of treatment
Arm/Group | Patients With PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 36 | 10 | 20
months | 22.1 [14.3 to NA] — The upper bounds of the confidence interval could not be calculated | 19.2 [9.2 to 19.2] | 10.2 [7.2 to 15.0]

20. Secondary Outcome: Median PFS on Last Prior Anti-cancer Therapy
Description: Progression Free Survival (PFS) is defined as the time in months from the start of treatment to the date of first documented disease progression or death due to any cause, which ever occurs first. PFS on last prior anti-cancer therapy is defined as the time in months from the start of last prior anti-cancer therapy to progression on that therapy.
Time Frame: Historical data collected at enrollment, all available data on prior therapy was collected
Population: Patients enrolled on any dose (Part 1 and Part 2) with data on progression-free survival for the most recent prior therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With a PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 45 | 51 | 142
months | 5.9 [4.2 to 8.3] | 31.0 [26.4 to 48.0] | 6.4 [4.3 to 8.3]

21. Secondary Outcome: Change From Baseline in Levels of KIT and PDGFRα Mutant Allele Fractions in Peripheral Blood
Description: Change of mutant allele fraction (MAF) summarizes the largest fold change. Change from baseline only displayed for patients with pre and post treatment MAF measurements. A positive number represents an increase in MAF. Data is only provided for patients that had both a baseline measurement and an end of treatment measurement.
Time Frame: Baseline and End of treatment
Population: Patients enrolled in Part 1 or Part 2 with a starting dose of 300 or 400 mg QD
Measure: Mean (Standard Deviation); unit: fraction of total
Groups:
- Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 mg or 400 mg QD: Part 1 and Part 2: Patients enrolled in Part 1 and Part 2 at a starting dose of 300 or 400 mg QD were included in the Part1/Part 2 safety and efficacy analysis.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
Arm/Group | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 mg or 400 mg QD
Number analyzed (Participants) | 1
fraction of total
  Change in PDGFRA MAF | 8.702 (NA) — Only one patient had data for this outcome measure so the standard deviation cannot be calculated
  Change in KIT MAF | 14.398 (NA) — Only one patient had data for this outcome measure so the standard deviation cannot be calculated

22. Secondary Outcome: KIT, PDGFRA, and Other Cancer-relevant Mutations Present in Tumor Tissue at Baseline and EOT
Description: Change in mutations in tumor tissue at baseline and end of treatment (EOT). EOT tumor biopsies were optional and there were no EOT samples collected.
Time Frame: Baseline and end of treatment
Population: Patients with pre-and post-treatment tumor biopsies. No patients provided a post-treatment biopsy.
Arm/Group | Patients With a PDGFRA D842V Mutation | 2L Patients Without a PDGFRA D842V Mutation | 3L Patients Without a PDGFRA D842V Mutation
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For each patient adverse event data were collected starting at the time of the first dose of study drug until 30 days after the final dose of study drug. Serious adverse event data were collected from the time the informed consent was signed until 30 days after the final dose of study drug. On average 8 months, up to 5 years.
Groups:
- Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD: Part 1: Patients received a starting dose of 200 mg QD for 28 days and they were assessed for dose limiting toxicities (DLT). If no DTLs were observed the dose escalation continued.
  Patients received avapritinib in continuous 28 day cycles until discontinuation.
Arm/Group | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD
All-Cause Mortality (participants affected / at risk) | 0/6 | 4/6 | 2/6 | 4/6 | 3/6 | 1/3 | 111/217
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 5/6 | 5/6 | 5/6 | 3/3 | 140/217
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/6 | 6/6 | 6/6 | 3/3 | 214/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD (N=3) | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD (N=217)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 8
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 8
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 7
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 18
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 6
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst rupture (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhagic cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dementia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 4
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to perineum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fistula discharge (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adrenal haemorrhage (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 30 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 60 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 90 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 135 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 200 mg QD (N=6) | Experimental: Part 1 Avapritinib (Formerly BLU-285) 600 mg QD (N=3) | Experimental: Part 1 and Part 2 Avapritinib (Formerly BLU-285) 300 or 400 mg QD (N=217)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 24
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 16
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 14
Periorbital oedema (Eye disorders) | 4 | 4 | 1 | 4 | 2 | 1 | 95
Lacrimation increased (Eye disorders) | 2 | 2 | 2 | 4 | 2 | 1 | 76
Eyelid oedema (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 18
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 14
Constipation (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 2 | 1 | 54
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0 | 4 | 0 | 1 | 36
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 22
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 22
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 18
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 16
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 11
Feeling cold (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 17
Influenza like illness (General disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 11
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 12
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 10
Blood bilirubin increased (Investigations) | 1 | 1 | 1 | 1 | 0 | 2 | 48
Weight decreased (Investigations) | 1 | 2 | 0 | 3 | 1 | 2 | 38
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 35
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 1 | 1 | 0 | 21
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 15
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 13
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 14
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 2 | 1 | 43
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 2 | 1 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1 | 1 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 14
Memory impairment (Nervous system disorders) | 2 | 2 | 0 | 2 | 2 | 1 | 73
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 2 | 2 | 2 | 51
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 3 | 1 | 2 | 40
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 16
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 13
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 11
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 3 | 1 | 1 | 32
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 20
Depression (Psychiatric disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 0 | 4 | 2 | 27
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 4 | 2 | 1 | 50
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 31
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 2 | 0 | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 13
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 2 | 3 | 2 | 3 | 88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT02508532/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT02508532/SAP_001.pdf